CLINICAL TRIAL: NCT07297693
Title: An Open-label, Randomized, Single-dose, Oral Administration, 2-sequence, 2-period, Crossover Study to Evaluate the Pharmacokinetics and Safety Between HIP2503 and HCP1306 in Healthy Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety Between HIP2503 and HCP1306 in Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-RIZE-101
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): * Period1 : HCP1306
  * Period2 : HIP2503
  Interventions: Drug: HIP2503; Drug: HCP1306
- Arm 2 (Experimental): * Period 1 : HIP2503
  * Period 2 : HCP1306
  Interventions: Drug: HIP2503; Drug: HCP1306

INTERVENTIONS:
Drug: HIP2503 — Take 1 orally disintegrating tablet once per period
Drug: HCP1306 — Take 1 tablet once per period

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic characteristics and safety between HIP2503 and HCP1306 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age 19~64 years in healthy volunteers
* 18 kg/m^2 ≤ BMI ≤ 30 kg/m^2, weight(men) ≥55kg / weight(women) ≥45kg
* Agrees that the person, spouse, or partner uses appropriate medically recognized contraception and does not provide sperm or eggs from the date of administration of the first investigational drug to 14 days after the administration of the last investigational drug
* Subjects who voluntarily decides to participate in this clinical trial and agree in writing to ensure compliance with the clinical trial

Exclusion Criteria:

* Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study
* Subjects who judged ineligible by the investigator

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-19 (Estimated); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
AUCt | 0~72 hours
  Pharmacokinetic evaluation
Cmax | 0~72 hours
  Pharmacokinetic evaluation

SECONDARY OUTCOMES:
Ka | 0~72 hours
  Pharmacokinetic evaluation
Concentration/Cmax_% | 0~72 hours
  Pharmacokinetic evaluation
AUCinf | 0~72 hours
  Pharmacokinetic evaluation
AUCt/AUCinf | 0~72 hours
  Pharmacokinetic evaluation
Tmax | 0~72 hours
  Pharmacokinetic evaluation
t1/2 | 0~72 hours
  Pharmacokinetic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Hee Ju Hong, Principal Investigator — H Plus Yangji Hospital
Locations (1):
- H plus Yangji Hospital, Seoul, Gwanak-gu, South Korea